CLINICAL TRIAL: NCT04269980
Title: Phentolamine Versus Magnesium Sulphate Infusion During Elective Lumbar Spine Surgery: a Randomized Double Blind Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, doaa rashwan, Assistant professor Doaa Rashwan, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMBSUREC/090222020/Ali
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Mean Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Care Provider)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (PHN) (Active Comparator): Group (PHN) (n=15): will receive hypotensive anesthesia with phentolamine infusion (Rogitamine, Egypharma) via syringe pump by adding 20 mg (2ml) of Phentolamine to 48 ml of normal saline making it to final concentration of 0.4 mg/ml at the rate of 0.1-2 mg/min according to the patients desired target blood pressure
  Interventions: Other: MAP
- Group MG (Active Comparator): Group MG (n=15): will receive hypotensive anesthesia with 40 mg/kg Magnesium sulphate as bolus in 15 min with infusion later on till end of surgery at the rate of 10 mg/kg/hr .
  Interventions: Other: MAP

INTERVENTIONS:
Other: MAP — MAP

SUMMARY:
The aim of this study is to evaluate the efficacy of controlled hypotensive anesthesia with phentolamine versus Magnesium sulfate in patients undergoing lumbar spine fusion surgery on blood loss, total dose of hypotensive agents and quality of surgical field.

DETAILED DESCRIPTION:
Patients and methods:

This study will be randomized controlled study ( RCT) and will be carried out in Beni-Suef University Hospital after the approval of institutional review board and ethical committee and obtaining a written informed consent from from ASA I and II patients undergoing elective lumbar spine surgery under general anesthesia. The primary outcome will be the achievement of controlled hypotension with MAP of 50-65 mmHg. The secondary outcomes will be blood loss, total dose of hypotensive agents and quality of surgical field.

This study will enroll 30 co-operative ASA physical status I & II patients of both sex aged 20-60 years undergoing elective lumbar spine surgry and study period will be 6 months.

Inclusion criteria:

orthopedic and neurological patients undergoing posterior lumbar spine fusion [American Society of Anesthesiologists (ASA) physical status 1 or 2, operation time of 3 to 5 h and mentally competent.

Exclusion Criteria:

1. operation time more than 5 h.
2. allergic reaction to drugs.
3. Patients with a history of liver, renal, heart and vascular failure, cardiac conduction disturbance.
4. opium addiction, any drug or substance abuse and chronic treatment with opium, non-steroidal anti-inflammatory drugs and calcium channel blockers (CCB).

The patients will be blinded to the study drugs and will be randomly assigned into two equal groups by opaque sealed envelope as follows:

Group (PHN) (n=15): will receive hypotensive anesthesia with phentolamine infusion (Rogitamine, Egypharma) via syringe pump by adding 20 mg (2ml) of Phentolamine to 48 ml of normal saline making it to final concentration of 0.4 mg/ml at the rate of 0.1-2 mg/min according to the patients desired target blood pressure.

Group MG (n=15): will receive hypotensive anesthesia with 40 mg/kg Magnesium sulphate as bolus in 15 min with infusion later on till end of surgery at the rate of 10 mg/kg/hr .

Anaesthetic technique:

On arrival to the operating room, standard monitoring will be established (pulse oximetry, electrocardiography, end-tidal carbon dioxide, and noninvasive arterial blood pressure monitoring), and oxygen will be delivered via a facemask. Two intravenous cannulas will placed; one (22 gauge) in a vein on the dorsum of the hand that the examined drug will be injected in and the other (20 gauge) in the opposite hand.

All patients will receive lactated ringer's solution at approximately 3-5 ml/kg/h perioperatively. The patients will be premedicated with Midazolam 0.05 mg/kg IV 3 minutes before induction. Anesthesia will induced by injecting 2.5 mg/kg propofol, 2 μg/kg fentanyl & 0.5 mg/kg atracurium.

The patients will be ventilated via face mask with 100 % oxygen at a rate of 4 L/min and isoflurane 1.2 %. After 3 minutes, the patients will be intubated using appropriate sized cuffed oral tube lubricated with lidocaine jelly 2 % , After induction of anesthesia, a radial arterial line from the non-dominant hand for continuous monitoring of mean arterial pressure (MAP) will be obtained.

Maintenance of anesthesia will done using isoflurane 1.2 % in 100 % O2. Muscle relaxation will be continued by atracurium 0.1 mg/kg every 20 min. All patients will be mechanically ventilated to maintain end-tidal carbon dioxide between 35-40 mmHg. For 5 minutes, no surgical interventions will be allowed in the subjects to assess target blood pressure.

The MAP will then gradually reduced in both groups to achieve and maintain the target MAP of 50-65 mmHg.

The surgical field will be evaluated by the surgeon using the 0-5 point bleeding scale (0: no bleeding, 1: low bleeding-bleeding does not require aspiration, 2: low bleeding-bleeding requires intermittent aspiration, 3: low bleeding-bleeding requires frequent aspiration, 4: moderate bleeding-bleeding becomes serious when aspirator is withdrawn from the surgical field, 5: serious bleeding-requires persistent aspiration, surgical field impossible) during the intra-operative period (13).

Patients who will develop severe hypotension (MAP <50 mmHg) will be managed by discontinuation of the hypotensive agent and reducing the concentration of isoflurane. If the MAP does not improve, 6 mg Ephedrine will be given IV & these patients will be excluded from the study. Patient who will develop bradycardia (<50 bpm) will be managed by intravenous atropine and will be then excluded from this study.

Infusion of the hypotensive agent will be stopped 5 minutes before the anticipated end of surgery. Any residual neuromuscular block will be antagonized with neostigmine 0.04 mg/kg and atropine 0.02 mg/kg IV.

The patients will be extubated on recovery of adequate tidal volume and sufficient respiratory efforts and transferred to recovery room for observation.

Surgeon's satisfaction will be recorded using the Likert technique or scale at the end of surgery (1 = very dissatisfied to 5 = completely satisfied).

The following data will be recorded :-

* Demographic data of the patients (Age, Sex, BMI) .
* MAP, HR, ETCO2 and SPO2 were recorded immediately prior to induction of anesthesia and subsequently every 5 min till the termination of anesthesia.
* Total phentolamine and magensium doses.
* The quality of surgical field will be evaluated by surgeon using the 0-5 point bleeding scale.
* The amount of blood loss will be determined by collecting the blood and rinsed fluid from the surgical field into the suction bottle by suctioning .The nurse who will not a part of the study made visual assessment of blood soaked gauge pieces that will be consumed during surgery.
* The time needed to reach the target blood pressure.
* Duration of surgery and anesthesia. HB and HTC preoperative and intraoperative Units of blood transfused
* In the recovery room, adverse effects such as nausea, vomiting, agitation, bradycardia, coughing, shivering, reflex tachycardia and rebound hypertension will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* orthopedic and neurological patients undergoing posterior lumbar spine fusion
* American Society of Anesthesiologists (ASA) physical status 1 or 2,
* operation time of 3 to 5 h
* mentally competent.

Exclusion Criteria:

* operation time more than 5 h.
* allergic reaction to drugs.
* Patients with a history of liver, renal, heart and vascular failure, cardiac conduction disturbance.
* opium addiction, any drug or substance abuse and chronic treatment with opium, non-steroidal anti-inflammatory drugs and calcium channel blockers (CCB).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
mean blood presure | intraopertaive

CONTACTS AND LOCATIONS:
Locations (1):
- Benisuef univercity, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided